CLINICAL TRIAL: NCT06864130
Title: The Alendronate Discontinuation Study
Brief Title: A Clinical Study on the Effect of Discontinuing Alendronate in Postmenopausal Women With Osteoporosis After a Treatment Period Without Fractures
Acronym: ALEXIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT 2023-510042-24; 2023-510042-24-01 (EU CTIS Number)
Record Dates: First submitted 2025-02-10; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis in Post-menopausal Women
Keywords: Alendronate; Discontinuation; Osteoporosis; Bone mineral density; post-menopausal
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Discontinuation of Alendronate (Experimental): Discontinuation of Alendronate treatment
  Interventions: Drug: Alendronate 70mg weekly
- Control group (No Intervention): The control group will continue Alendronate treatment, but shift to project-sponsored product (70 mg Alendronate weekly)

INTERVENTIONS:
Drug: Alendronate 70mg weekly — The intervention is discontinuation of Alendronate
  Arms: Discontinuation of Alendronate

SUMMARY:
The goal of this clinical trial is to study the effects of discontinuation of Alendronate treatment for three years. The participants are postmenopausal women with osteoporosis, who have had a treatment period without fractures. The study will answer:

* What is the rate of fragility fractures during the study? The hypothesis is that discontinuation of Alendronate after a fracture-free period does not raise the 3-year fracture risk.
* Are there predictors of significant bone loss after discontinuation of Alendronate? The hypothesis is that clinical, biochemical, cellular, or molecular characteristics can predict bone loss.

Researchers will compare the outcomes of discontinuation of Alendronate with continuing treatment. Participants will be randomly assigned to a group.

Participants will:

* Either take alendronate once weekly for three years OR discontinue their treatment
* Visit the clinic at 6 and 18 months for blood samples
* Visit the clinic at the start of the study and after 1, 2, and 3 years for bone scans and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Postmenopausal
* Current treatment with Alendronate
* Alendronate treatment >3 år AND no fracture OR
* Alendronate treatment >5 år AND latest low energy fracture > 3 years ago

Exclusion Criteria:

* T-score < - 3,5 in hip (total hip or femoral neck) or lumbar spine
* Treatment with systemic glucocorticoids, ongoing or within 12 months
* Uncontrolled inflammatory disease
* Active malignancy
* eGFR < 40 mL/min
* Atypical femur fracture (ever)
* OsteoNecrosis of the Jaw (active)
* Unable to give inform consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only biological females will be enrolled.
Enrollment: 1400 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-09-15 (Estimated)

PRIMARY OUTCOMES:
Fragility fractures | From enrollment to the end of the 3 year study period.
  Incidence of fragility fractures during the study period

SECONDARY OUTCOMES:
Changes in bone mineral density (BMD) | Baseline, 12, 24 and 36 months
  Changes in lumbar spine and total hip BMD measured by dual energy X-ray arbsorptiometry. The three follow-up scans will be analyzed by a technician blinded to participant allocation, ie this person will not meet the patient and the patient will not be able see the results of the scans until the final study visit.
Bone turn over marker (CTX) | Blood samples are performed at baseline, 6, 12, 18, 24, and 36 months.
  Fasting blood samples will be performed during the study period to analyze changes in carboxy-terminal collagen crosslinks (CTX).
Bone turn over marker (P1NP) | Blood samples are performed at baseline, 6, 12, 18, 24, and 36 months.
  Fasting blood samples will be performed during the study period to analyze changes in procollagen type I N-terminal propeptide (PINP).
Restart Criteria | From enrollment to the end of the study period at 3 years
  The proportion of participants meeting restart criteria during the study period. Restart criteria is defined as: Participants experiencing boneloss exceeding 10% from baseline in any region, one clinical vertebral fracture, two low energy fractures (including morphometric vertebral fracture but excluding fractures of scull, fingers or toes) are withdrawn from the study and offered treatment with alendronate or zoledronic acid after new diagnostic work-up.
Adverse Events | From enrollment to the end of the 3 year study period.
  At baseline a thoroughly physical examination of the participants and questioning concerning any conditions or diseases will take place. This way the investigators will be able to evaluate possible changes throughout the study. Patients will be interviewed about the occurrence of AEs at each visit from the first trial related activity after the subject has signed the informed consent. Subjects that experience adverse events or develop a disease during the trial period will be managed until the condition is cured or stationary. If this is not the case at the end of the study, subjects will be referred to a relevant physician, e.g. the general practitioner or a specialist, to be followed up.

OTHER OUTCOMES:
Osteoclastassay | Baseline and 12 months
  Osteoclasts differentiation, formation, activity and response to Alendronate in cultures derived from peripheal blood at baseline and 12 months, from a subgroup of 35 from each arm (70 participants in total).
Molecular bone histology | 12 and 36 months
  Iliac crest bone biopsy specimens will be obtained to evaluate the effect of discontinuation of alendronate on cortical and trabecular bone resorption and formation by histomorphometry. These results will be compared with results of bone turnover markers. Biopsies will be obtained of maximum 35 from each treatment group at 12 and 36 months (in totalt 140 participants).
Epigenetic analysis | Baseline
  Epigenetic analysis of peripheal blood with focus on the degree of methylation.

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Hermann, MD, PhD., Principal Investigator — Odense Universitetshospital / Odense University Hospital
Locations (7):
- Denmark (7):
  - Aalborg University Hospital, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Esbjerg Og Grindsted Sygehus, Esbjerg
  - Copenhagen University Hospital (Herlev), Herlev
  - Nordsjaellands Hospital (Hillerød), Hillerød
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No